CLINICAL TRIAL: NCT01268631
Title: Mechanism-based Choice of Therapy: Can Treatments Success in Fibromyalgia Patients be Coupled to Psychophysical Pain Modulation Profile?
Acronym: MTF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: University of California, Davis (Other); Rambam Health Care Campus (Other)
Responsible Party: Jacob Ablin, MD, Director Fibromyalgia clinic, Tel Aviv Sourasky Medical Center, Tel Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0368-10-TLV
Record Dates: First submitted 2010-12-29; First posted 2010-12-31 (Estimated); Last update posted 2010-12-31 (Estimated); Status verified 2010-12

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Pain modulation
MeSH Terms: conditions — Fibromyalgia | interventions — Duloxetine Hydrochloride; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine (Active Comparator): Initial dose of 30 mg/d will be given for one week, in order to minimize possible side effects and drop outs, and then a fixed dose of 60 mg/d will be given for additional 4 weeks. The assessing person will contact patients by phone every week during the treatment period to receive the pain score for the last 24 hours, so we will have an indication of the effect among patients will discontinue medication. Patients will be asked to visit the clinic during the last week of treatment, for assessment of clinical pain (questionnaires) and pain modulation.
  Interventions: Drug: Duloxetine; Drug: Pregabalin
- Pregabalin (Active Comparator): Initial dose of 75x2mg/d for one week, and then fixed dose of 150x2mg/d for the following 4 weeks. Drug should not be taken with meals. Same protocol will be applied as for Duloxetine.
  Interventions: Drug: Duloxetine; Drug: Pregabalin

INTERVENTIONS:
Drug: Duloxetine — Initial dose of 30 mg/d will be given for one week, in order to minimize possible side effects and drop outs, and then a fixed dose of 60 mg/d will be given for additional 4 weeks. The assessing person will contact patients by phone every week during the treatment period to receive the pain score for the last 24 hours, so we will have an indication of the effect among patients will discontinue medication. Patients will be asked to visit the clinic during the last week of treatment, for assessment of clinical pain (questionnaires) and pain modulation.
Drug: Pregabalin — Initial dose of 75x2mg/d for one week, and then fixed dose of 150x2mg/d for the following 4 weeks. Drug should not be taken with meals. Same protocol will be applied as for Duloxetine.

SUMMARY:
Hypothesis:

Response to therapy in fibromyalgia can be improved by coupling of specific medications to the individual patterns of dysfunctional pain modulation. Individuals exhibit wide range of pain modulating capabilities that can be assessed by dynamic psychophysical testing. Those that exhibit less efficient endogenous analgesia and/or increased pain summation are known to be more prone to suffer from pain. Tailoring medications to compensate for the specific dysfunctioning modulatory mechanism will improve pain control.

DETAILED DESCRIPTION:
Plan Overview:

The study will be conducted as a double - blind research. After undergoing evaluation of pain processing as detailed in the protocol, patients recruited will be randomised to receive Douloxetine or Pregabalin, two medications with evidence - based efficacy in the treatment of the fibromyalgia syndrome. After the first week of the study, all patients recruited will receive active treatment with one of these two medications.

This project will recruit fibromyalgia patients. Those patients will be treated with either Duloxetine or Pregabalin, and follow up will be made on the response to treatment as well as for possible change in pain modulation.

Study population:

We plan that 40 fibromyalgia patients will complete the analgesic treatment phase for each of the two medications. Considering an expected drop out of 30-50%, 150 patients will be recruited.

Inclusion criteria: fibromyalgia patients. All patients will undergo physical examination and tender point evaluation to ascertain fulfillment of the ACR 1990 criteria for classification of fibromyalgia (Wolfe et al 1990) i.e. the presence of widespread pain lasting at least 3 months and the presence of tenderness in at least 11 of 18 tender points.

Exclusion criteria: age below 18 and above 80; patients with cognitive dysfunction precluding use of psychophysics, those who cannot communicate in Hebrew, abnormal renal function with creatinine above 1.5, and elevated liver enzymes >x3 upper limit. Since the duloxetine has the potential to act as both substrate and an inhibitor of cytochrome P4502D6 (CYP2D6) inhibiting, caution should be used when other CYP2D6 substrates and inhibitors (some tricyclic antidepressants and SSRIs) are coadministered with duloxetine (Skinner et al., 2003). Patients currently treated with Douloxetine, Pregabalin, Gabapentin, Milnacipran, amitryptiline or other SSRIs, NSRIs or tricyclic medications will not be recruited unless they consent to discontinue prior medications for three weeks before enrolment to the study. During this period the use of NSAIDS and common analgesic medication will be permitted.

Patietns not currently treated with such medications can be recruited. Patietns suffering from chronic pain due to a known active malignancy or other localized cause (e.g. fracture, Herpes Zoster etc.) will not be recruited.

Systemic pain modulation:

1. DNIC will be assessed as the difference of pain ratings to 'test stimulus' applied before and during the immersion of the contralateral hand into hot water bath ('conditioning stimulus'). 'Test stimulus' is a 30" contact heat stimulus (30x30 mm2 thermode, TSA-2001, Medoc) delivered on the non-dominant forearm at the individually-predetermined temperature that evoked pain intensity of 60 in a 0-100 NPS (more details in Granot et al., 2006). The stimulus temperature will rise at 2oC/sec from 32oC to the destination temperature. Fifteen minutes after the completion the first pre-immersion test, patient will be asked to immerse his/her dominant hand for 1' into the water bath of 46.5oC (Heto Cooling Bath CBN 8-30, Allerod, Denemark), while second application of the 'test stimulus' will be repeated during last 30" of immersion. To assess the residual DNIC effect 3' after end of immersion, the 'test stimulus' will be applied for the third time. During each application of 'test stimulus' patient will be asked to rate his thermal pain intensity every 10' (NPS, 4 readings total).
2. Mechanical Temporal Summation (TS) will be assessed by the 6.45mN von Frey filament (Stoeteling Ltd. US). A single stimulus, and then a train of 10 successive stimuli will be applied to the volar forearm, with ISI of 1". Pricking pain scores (0-100 on NPS) will be obtained after the single, and then at the end of the train. The difference between these scores will be calculated as TS.

Static pain pyschophysics:

1. Sensory mechanical tactile thresholds will be determined using von Frey filaments, on the volar forearm. Stimuli ascending from lowest filament, until subject reports about clear tactile sensation in 2/3 applications.
2. Sensory thermal thresholds will be determined using TSA, on the volar forearm. Temperature will increase or decrease and the patient will be asked to press a button when he perceives the temperature as warm or cold, respectively.
3. Mechanical pain threshold will be assessed similar to above, starting at von Frey of 4.88mN on the volar forearm.
4. Pain thermal thresholds will be determined using TSA, on the volar forearm. Temperature will increase or decrease and the patient will be asked to press a button when he perceives the temperature as painful.

3.2.4.4. Clinical pain assessment Mean and maximal pain scores during the last week will be obtained from subjects at each test session. Characteristics of pain will be assessed using the validated Hebrew version of the Fibromyalgia Impact questionnaire (FIQ) (Buskila et al 1996).

In addition, intensity and level of pain interfering with life will be assessed using the Brief Pain Inventory (BPI) (Cleeland & Ryan, 1994) as well as the pain catastrophizing level and the Spielberger state and trait anxiety inventory questionnaire. The Pittsburgh sleep quality index (PSQI) will also be assessed. The records of use of analgesic and other treatments, including use of opioids will be obtained.

Pain relief treatments:

Our previous experience indicates that even within the chronic pain patients there is still a wide enough range of DNIC and TS. Treatments will be given for 6 weeks, where the physician administering the treatment will not know what treatment is given (code can be broken at any stage for serious adverse events at the discretion of the PI). Thus both patients and assessing personal will be blinded to type to therapy. In order to evaluate the placebo effect, for all patients, the first week of treatment will be the administration of non-active placebo. All patients will proceed to the active treatment stage, but those reporting 50% or more pain reduction after placebo treatment will be analyzed separately. Some of the patients, in addition to the described lab tests schedule, will be invited and tested for their experimental pain perception at the end of the placebo period. For the purpose of blinding across the treatments, every medication will be administered twice daily (using different capsule colors for the morning and evening tablets). The use of rescue pain alleviation by NSAIDs will be permitted at any stage.

a. Duloxetine. Initial dose of 30 mg/d will be given for one week, in order to minimize possible side effects and drop outs, and then a fixed dose of 60 mg/d will be given for additional 4 weeks. The assessing person will contact patients by phone every week during the treatment period to receive the pain score for the last 24 hours, so we will have an indication of the effect among patients will discontinue medication. Patients will be asked to visit the clinic during the last week of treatment, for assessment of clinical pain (questionnaires) and pain modulation.

Outcome measures and data analysis The primary outcome is the correlations between pain modulation and drug effect. This will be explored for each stage, and in relation to clinical pain and the other pain variables such as hyperalgesia. Logistic regression models will be constructed to best predict drugs effect considering modulation mechanisms, time of measurement, acute and chronic pain. NNTs will be calculated based on the modulation state of the patients (>50% pain relief will be considered as successful treatment).

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia patients. All patients will undergo physical examination and tender point evaluation to ascertain fulfillment of the ACR 1990 criteria for classification of fibromyalgia (Wolfe et al 1990) i.e. the presence of widespread pain lasting at least 3 months and the presence of tenderness in at least 11 of 18 tender points.

Exclusion Criteria:

* Age below 18 and above 80
* Patients with cognitive dysfunction precluding use of psychophysics, those who cannot communicate in Hebrew, abnormal renal function with creatinine above 1.5, and elevated liver enzymes >x3 upper limit. Since the duloxetine has the potential to act as both substrate and an inhibitor of cytochrome P4502D6 (CYP2D6) inhibiting, caution should be used when other CYP2D6 substrates and inhibitors (some tricyclic antidepressants and SSRIs) are coadministered with duloxetine (Skinner et al., 2003). Patients currently treated with Douloxetine, Pregabalin, Gabapentin, Milnacipran, amitryptiline or other SSRIs, NSRIs or tricyclic medications will not be recruited unless they consent to discontinue prior medications for three weeks before enrolment to the study. During this period the use of NSAIDS and common analgesic medication will be permitted.
* Patients not currently treated with such medications can be recruited.
* Patients suffering from chronic pain due to a known active malignancy or other localized cause (e.g. fracture, Herpes Zoster etc.) will not be recruited.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
correlations between pain modulation and drug effect | 2 years
  This will be explored for each stage, and in relation to clinical pain and the other pain variables such as hyperalgesia

CONTACTS AND LOCATIONS:
Locations (1):
- Rheumatology Institute, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Granot M, Granovsky Y, Sprecher E, Nir RR, Yarnitsky D. Contact heat-evoked temporal summation: tonic versus repetitive-phasic stimulation. Pain. 2006 Jun;122(3):295-305. doi: 10.1016/j.pain.2006.02.003. Epub 2006 Mar 15. PMID 16540248
- [Background] Skinner MH, Kuan HY, Pan A, Sathirakul K, Knadler MP, Gonzales CR, Yeo KP, Reddy S, Lim M, Ayan-Oshodi M, Wise SD. Duloxetine is both an inhibitor and a substrate of cytochrome P4502D6 in healthy volunteers. Clin Pharmacol Ther. 2003 Mar;73(3):170-7. doi: 10.1067/mcp.2003.28. PMID 12621382
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- [Background] Buskila D, Neumann L. Assessing functional disability and health status of women with fibromyalgia: validation of a Hebrew version of the Fibromyalgia Impact Questionnaire. J Rheumatol. 1996 May;23(5):903-6. PMID 8724306